CLINICAL TRIAL: NCT03507933
Title: Evaluation of the Effectiveness of Surgical Treatment of Villo-nodular Synovitis of the Hip in Children in a Retrospective Case Series
Brief Title: Evaluation of the Effectiveness of Surgical Treatment of Villo-nodular Synovitis of the Hip in Children
Acronym: SVN
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Lille Catholic University (Other)
Responsible Party: Sponsor
Other Study IDs: OBS-0033
Record Dates: First submitted 2018-03-07; First posted 2018-04-25 (Actual); Last update posted 2018-04-25 (Actual); Status verified 2018-03

CONDITIONS: Synovitis
Keywords: villo-nodular synovitis; Hip; Surgery
MeSH Terms: conditions — Synovitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Villo-nodular synovitis can affect the joints, bursae or tendon sheaths. This condition is rare, with 1.8 cases per million inhabitants. The hip is affected in 3.6 to 18.1% of cases. The age of predilection is between 30 and 50 years old and this condition is rarely described in children.

Two articles report a case of villous-nodular synovitis of the child's hip. Surgical treatment by resection seems to be consensus but various adjuvant treatments are also proposed. A case of villous-nodular synovitis of the hip in children was treated without surgical intervention. The main objective of this study was to evaluate the efficacy of surgical treatment of villous nodular synovitis of the hip in children.

DETAILED DESCRIPTION:
French multicentric cases serie

ELIGIBILITY:
Inclusion Criteria:

* Children with histologically villo-nodular synovitis of the hip
* Surgical procedures performed for the treatment of this synovitis

Exclusion Criteria:

* Degree of bone maturation and Risser test greater than 4 at the time of diagnosis
* Parents opposing the use of their child's data / Patient opposing the use of his/her data

Ages: 10 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Children operated for villo-nodular synovitis of the hip
Sampling Method: Non-Probability Sample
Enrollment: 6 (Estimated)
Dates: Start 2018-01-30 (Actual); Primary Completion 2018-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in the range of motion of the hip in degrees | before surgery and 4 months after surgery
  Evaluation of extension / flexion / abduction / adduction / external rotation / internal rotation of the hip
Incidence of signal changes in the X-Ray | 4 months after surgery
Incidence of signal changes in the MRI | 4 months after surgery

SECONDARY OUTCOMES:
Change from baseline in the scale measure of patient's pain intensity | before surgery and 4 months after surgery
Incidence of complications after surgery | 4 month after surgery
Number of additional treatments used in addition to surgery | 4 month after surgery
  Frequency of adjuvant treatments
Change from baseline in the physical activity evaluated by a questionnaire | before surgery and 4 months after surgery
  yes /no questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Raphael Coursier, MD, Principal Investigator — Lille Catholic University
Locations (1):
- Lille Catholic University, Lille, France